CLINICAL TRIAL: NCT02023099
Title: A Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) in Treatment-Naïve and Treatment-Experienced Japanese Adults With Subgenotype 1b Chronic Hepatitis C Virus (HCV) Infection With and Without Compensated Cirrhosis (GIFT I)
Brief Title: Study to Evaluate the Efficacy and Safety of ABT-450/Ritonavir/ABT-267 (ABT-450/r/ABT-267) in Japanese Adults With Subgenotype 1b Chronic Hepatitis C Virus (HCV) Infection
Acronym: GIFT I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-004
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2016-09

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C; Genotype 1b; Cirrhotic; Treatment Experienced; Treatment Naive; Japanese; ombitasvir; paritaprevir; ritonavir; VIEKIRAX Combination Tablets
MeSH Terms: conditions — Hepatitis C | interventions — ombitasvir; paritaprevir; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Substudy 1, Arm A: DB 2-DAA (Experimental): Double-blind (DB) 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2 direct-acting antiviral agents [2-DAA]) once daily (QD) for 12 weeks in participants without cirrhosis
  Interventions: Drug: ABT-450/r/ABT-267
- Substudy 1, Arm B: DB Placebo, Followed by OL 2-DAA (Placebo Comparator): DB placebo QD for 12 weeks followed by open-label (OL) 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2-DAA) QD for 12 weeks in participants without cirrhosis
  Interventions: Drug: ABT-450/r/ABT-267; Drug: Placebo
- Substudy 2, Arm C: OL 2-DAA (Experimental): OL 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2-DAA) QD for 12 weeks in participants with compensated cirrhosis
  Interventions: Drug: ABT-450/r/ABT-267

INTERVENTIONS:
Drug: ABT-450/r/ABT-267 — Tablet; ABT-450 coformulated with ritonavir and ABT-267
  Other Names: ABT-267 also known as ombitasvir; ABT-450 also known as paritaprevir; ritonavir also known as Norvir; VIEKIRAX Combination Tablets; Qurevo; Technivie; VIEKIRA Combination Tablets
Drug: Placebo — Tablet
  Arms: Substudy 1, Arm B: DB Placebo, Followed by OL 2-DAA

SUMMARY:
This is a phase 3, double-blinded, multicenter study. The study will consist of 2 substudies: Substudy 1 (SS1) will be double-blinded and enroll non-cirrhotic subjects and Substudy 2 (SS2) will be open label and enroll subjects with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV-infection prior to study enrollment
* Screening laboratory result indicating HCV subgenotype 1b infection
* Subject has plasma HCV RNA level greater than 10,000 IU/mL at Screening
* Voluntarily sign an informed consent
* Females must be practicing specific forms of birth control on study treatment, or be post-menopausal for more than 2 years or surgically sterile

Exclusion Criteria:

* Co-infection of Hepatitis B Virus (HBV), human immunodeficiency virus (HIV) or any HCV genotype other than subgenotype 1b
* Prior therapy with direct acting antiviral agents for the treatment of HCV, including telaprevir, simeprevir and boceprevir
* Any cause of liver disease other than chronic HCV-infection, including but not limited to the following: hemochromatosis; alpha-1 antitrypsin deficiency; Wilson's disease; autoimmune hepatitis; alcoholic liver disease; drug-related liver disease; clinically significant laboratory abnormalities; uncontrolled clinically significant disease, disorder or medical illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nori Yachi, Study Director — AbbVie

REFERENCES:
- [Result] Kumada H, Chayama K, Rodrigues L Jr, Suzuki F, Ikeda K, Toyoda H, Sato K, Karino Y, Matsuzaki Y, Kioka K, Setze C, Pilot-Matias T, Patwardhan M, Vilchez RA, Burroughs M, Redman R. Randomized phase 3 trial of ombitasvir/paritaprevir/ritonavir for hepatitis C virus genotype 1b-infected Japanese patients with or without cirrhosis. Hepatology. 2015 Oct;62(4):1037-46. doi: 10.1002/hep.27972. Epub 2015 Aug 25. PMID 26147154
- [Derived] Gopalakrishnan S, Khatri A, Mensing S, Redman R, Menon R, Zha J. Exposure-Response Relationship for Ombitasvir and Paritaprevir/Ritonavir in Hepatitis C Virus Subgenotype 1b-Infected Japanese Patients in the Phase 3 Randomized GIFT-I Study. Adv Ther. 2016 Apr;33(4):670-83. doi: 10.1007/s12325-016-0320-y. Epub 2016 Mar 21. PMID 27084721
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Substudy 1, Arm A: DB 2-DAA | Substudy 1, Arm B: DB Placebo, Followed by OL 2-DAA | Substudy 2, Arm C: OL 2-DAA
Started | 215 | 106 | 42
Completed | 212 | 106 | 39
Not Completed | 3 | 0 | 3
Not completed — Non-fatal Adverse Event (AE) | 0 | 0 | 1
Not completed — Withdrawn Consent | 3 | 0 | 1
Not completed — Non-treatment-emergent Fatal AE | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Substudy 1, Arm A: DB 2-DAA: DB 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2-DAA) QD for 12 weeks in participants without cirrhosis
- Substudy 1, Arm B: DB Placebo, Followed by OL 2-DAA: DB placebo QD for 12 weeks followed by OL 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2-DAA) QD for 12 weeks in participants without cirrhosis
- Total: Total of all reporting groups
Arm/Group | Substudy 1, Arm A: DB 2-DAA | Substudy 1, Arm B: DB Placebo, Followed by OL 2-DAA | Substudy 2, Arm C: OL 2-DAA | Total
Number analyzed (Participants) | 215 | 106 | 42 | 363
Age, Customized [Number; unit: participants]
  < 65 years | 129 | 59 | 21 | 209
  ≥ 65 years | 86 | 47 | 21 | 154
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 59 | 22 | 216
  Male | 80 | 47 | 20 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Non-cirrhotic Treatment-Naïve Participants Who Are Eligible for Interferon (IFN)-Based Therapy and Who Have High Viral Load in the DB Active Treatment Group With a Sustained Virologic Response 12 Weeks Post-treatment
Description: The percentage noncirrhotic treatment-naïve participants who were eligible for IFN-based therapy and who had high viral load at baseline (HCV RNA ≥ 100,000 IU/mL) in the DB active treatment group with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of active study drug (SVR12). Among noncirrhotic treatment-naïve participants who were eligible for IFN-based therapy and who had high viral load at baseline, superiority of Arm A to a clinically relevant threshold based on historical SVR rate with telaprevir plus pegylated interferon alpha/ribavirin (pegIFN/RBV) in treatment-naïve, non-cirrhotic patients with high viral load; the lower bound of 95% confidence interval (LCB) had to exceed 63% to achieve superiority. The 95% confidence interval was calculated using the normal approximation to the binomial distribution.
Time Frame: 12 weeks after the last dose of study drug
Population: Primary Efficacy Population: randomized non-cirrhotic treatment-naïve participants who are eligible for interferon-based therapy and who have high viral load and received at least one dose of double-blind ABT-450/r/ABT-267.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA
Number analyzed (Participants) | 112
percentage of participants | 94.6 [90.5 to 98.8]

2. Secondary Outcome: Percentage of Participants in the Active Treatment Group With On-treatment Virologic Failure During Treatment
Description: On-treatment virologic failure among all randomized non-cirrhotic participants who received at least one dose of DB ABT-450/r/ABT-267 and all enrolled participants with compensated cirrhosis who received at least one dose of OL ABT-450/r/ABT-267. On-treatment virologic failure is defined as the occurrence of at least one of the following:
  * confirmed HCV RNA ≥ LLOQ (defined as 2 consecutive HCV RNA measurements ≥ LLOQ) at any point during treatment after HCV RNA < LLOQ (rebound), or
  * confirmed increase from nadir in HCV RNA (defined as 2 consecutive HCV RNA measurements > 1 log10 IU/mL above nadir) at any time point during treatment (rebound), or
  * HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks (≥ 36 days) of treatment (failure to suppress).
  The 95% confidence interval was calculated using the Wilson's score method.
Time Frame: up to 12 weeks
Population: Intent-to-treat (ITT) population: randomized/enrolled participants who received at least 1 dose of DB study drugs in Substudy 1 (Substudy 1 ITT population) and completed treatment; n=number of participants in the given subpopulation (among noncirrhotic participants, a single participant could potentially be included in more than 1 subpopulation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA | Substudy 2, Arm C: OL 2-DAA
Number analyzed (Participants) | 215 | 42
percentage of participants | 0.5 [0.1 to 2.6] | 2.4 [0.4 to 12.3]

3. Secondary Outcome: Percentage of Participants in the Substudy 1 Arm A Active Treatment Group With On-treatment Virologic Failure During Treatment, by Subpopulation
Description: On-treatment virologic failure among all randomized non-cirrhotic participants who received at least one dose of DB ABT-450/r/ABT-267 in the following subpopulations: noncirrhotic treatment-naïve (T-naïve) participants with a high baseline (BL) viral load (HCV RNA ≥ 100,000 IU/mL) who are eligible for IFN-based therapy (IFN-BT), a low viral load (HCV RNA < 100,000 IU/mL), or who are ineligible for IFN-BT; noncirrhotic treatment-experienced (T-exp) participants who relapsed after prior IFN-BT, who were nonresponders to prior IFN-BT, or who were intolerant to IFN-BT. On-treatment virologic failure is defined in Outcome measure 2. The 95% confidence interval was calculated using the Wilson's score method.
Time Frame: up to 12 weeks
Population: ITT population: all randomized/enrolled participants who received at least 1 dose of active DB study drugs in Substudy 1 (Substudy 1 ITT population, Arm A).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA
Number analyzed (Participants) | 215
percentage of participants
  T-naïve: high BL viral load, IFN-eligible; n=112 | 0 [0.0 to 3.3]
  T-naïve: low BL viral load; n=6 | 0 [0.0 to 39.0]
  T-naïve: IFN-ineligible; n=23 | 0 [0.0 to 14.3]
  T-exp. w/prior IFN-BT: relapser; n=22 | 0 [0.0 to 14.9]
  T-exp. w/prior IFN-BT: nonresponder; n=28 | 0 [0.0 to 12.1]
  T-exp. w/prior IFN-BT: IFN-intolerant; n=26 | 3.8 [0.7 to 18.9]

4. Secondary Outcome: Percentage of Participants in the Active Treatment Group With Post-treatment Relapse
Description: Post-treatment relapse among all randomized non-cirrhotic participants who received at least one dose of DB ABT-450/r/ABT-267 and completed treatment, and all enrolled participants with compensated cirrhosis who received at least one dose of OL ABT-450/r/ABT-267 and completed treatment. Relapse was defined as confirmed HCV RNA ≥ LLOQ (defined as 2 consecutive HCV RNA measurements ≥ LLOQ) between the final treatment visit and 12 weeks after the last dose of study drugs among participants completing treatment and with HCV RNA < LLOQ at the final treatment visit and at least one post-treatment HCV RNA value. The 95% confidence interval was calculated using the Wilson's score method.
Time Frame: within 12 weeks after last dose of study drug
Population: ITT population: all randomized/enrolled participants who received at least 1 dose of active DB study drugs in Substudy 1 (Substudy 1 ITT population, Arm A) or at least 1 dose of OL study drugs in Substudy 2 (Substudy 2 ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA | Substudy 2, Arm C: OL 2-DAA
Number analyzed (Participants) | 209 | 40
percentage of participants | 2.4 [1.0 to 5.5] | 5.0 [1.4 to 16.5]

5. Secondary Outcome: Percentage of Participants in Substudy 1 Arm A Active Treatment Group With Post-treatment Relapse, by Subpopulation
Description: Post-treatment relapse among all randomized non-cirrhotic participants who received at least one dose of DB ABT-450/r/ABT-267 and completed treatment, in the following subpopulations: noncirrhotic treatment-naïve (T-naïve) participants with a high baseline (BL) viral load (HCV RNA ≥ 100,000 IU/mL) who are eligible for IFN-based therapy (IFN-BT), a low BL viral load (HCV RNA < 100,000 IU/mL), or who are ineligible for IFN-BT; noncirrhotic treatment-experienced (T-exp) participants who relapsed after prior IFN-BT, who were nonresponders to prior IFN-BT, or who were intolerant to IFN-BT.
  Relapse was defined as confirmed HCV RNA ≥ LLOQ (defined as 2 consecutive HCV RNA measurements ≥ LLOQ) between the final treatment visit and 12 weeks after the last dose of study drugs among participants completing treatment and with HCV RNA < LLOQ at the final treatment visit and at least one post-treatment HCV RNA value. The 95% confidence interval was calculated using the Wilson's score method.
Time Frame: within 12 weeks after last dose of study drug
Population: ITT population: all randomized/enrolled participants who received at least 1 dose of active DB study drugs in Substudy 1 (Substudy 1 ITT population, Arm A) and completed treatment; n=number of participants in the given subpopulation (among noncirrhotic participants, a single participant could potentially be included in more than 1 subpopulation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA
Number analyzed (Participants) | 209
percentage of participants
  T-naïve: high BL viral load, IFN-eligible; n=109 | 2.8 [0.9 to 7.8]
  T-naïve: low BL viral load; n=6 | 0 [0 to 39.0]
  T-naïve: IFN-ineligible; n=22 | 4.5 [0.8 to 21.8]
  T-exp. w/prior IFN-BT: relapser; n=21 | 0 [0 to 15.5]
  T-exp. w/prior IFN-BT: nonresponder; n=28 | 0 [0 to 12.1]
  T-exp. w/prior IFN-BT: IFN-intolerant; n=25 | 4.0 [0.7 to 19.5]

6. Secondary Outcome: Percentage of Participants in the Active Treatment Group With Sustained Virologic Response 12 Weeks Post-treatment
Description: Sustained virologic response (plasma HCV RNA level < LLOQ) 12 weeks after the last dose of study drug for all randomized non-cirrhotic participants who received at least one dose of DB ABT-450/r/ABT-267 and for all enrolled participants with compensated cirrhosis who received at least one dose of open-label ABT-450/r/ABT-267. The 95% confidence interval was calculated using the Wilson's score method.
Time Frame: 12 weeks after last dose of study drug
Population: ITT population: all randomized/enrolled participants who received at least 1 dose of DB study drugs in Substudy 1 (Substudy 1 ITT population) or at least 1 dose of OL study drugs in Substudy 2 (Substudy 2 ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA | Substudy 2, Arm C: OL 2-DAA
Number analyzed (Participants) | 215 | 42
percentage of participants | 94.9 [91.1 to 97.1] | 90.5 [77.9 to 96.2]

7. Secondary Outcome: Percentage of Participants in Substudy 1 Arm A Active Treatment Group With Sustained Virologic Response 12 Weeks Post-Treatment, by Subpopulation
Description: Sustained virologic response (plasma HCV RNA level < LLOQ) 12 weeks after the last dose of study drug for all randomized non-cirrhotic participants who received at least one dose of DB ABT-450/r/ABT-267 in the following subpopulations: noncirrhotic T-naïve participants with a high BL viral load (HCV RNA ≥ 100,000 IU/mL) who are eligible for IFN-BT; noncirrhotic T-naïve participants with low BL viral load (HCV RNA < 100,000 IU/mL); noncirrhotic T-naïve participants who are ineligible for IFN-BT; noncirrhotic T-exp participants who relapsed after prior IFN-BT; noncirrhotic T-exp participants who were nonresponders to prior IFN-BT; noncirrhotic T-exp participants who were intolerant to IFN-BT. The 95% confidence interval was calculated using the Wilson's score method.
Time Frame: 12 weeks after last dose of study drug
Population: ITT population: all randomized/enrolled participants who received at least 1 dose of active DB study drugs in Substudy 1 (Substudy 1 ITT population, Arm A); n=number of participants in the given subpopulation (among noncirrhotic participants, a single participant could potentially be included in more than 1 subpopulation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1, Arm A: DB 2-DAA
Number analyzed (Participants) | 215
percentage of participants
  T-naïve: all; n=139 | 94.2 [89.1 to 97.1]
  T-naïve: high BL viral load, IFN-eligible; n=112 | 94.6 [88.8 to 97.5]
  T-naïve: low BL viral load; n=6 | 100 [61.0 to 100]
  T-naïve: IFN-ineligible; n=23 | 91.3 [73.2 to 97.6]
  T-exp. w/prior IFN-BT: all; n=76 | 96.1 [89.0 to 98.6]
  T-exp. w/prior IFN-BT: relapser; n=22 | 95.5 [78.2 to 99.2]
  T-exp. w/prior IFN-BT: nonresponder; n=28 | 100 [87.9 to 100]
  T-exp. w/prior IFN-BT: IFN-intolerant; n=26 | 92.3 [75.9 to 97.9]

ADVERSE EVENTS:
Time Frame: AEs collected from time of informed consent through 30 days post-study drug dosing (dosing period was 12 or 24 weeks [12 weeks of placebo followed by 12 weeks of DAAs]); Serious AEs collected up to post-treatment Week 48.
Groups:
- Substudy 1, Arm A: DB 2-DAA: DB 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2 direct-acting antiviral agents [2-DAA]) once daily (QD) for 12 weeks in participants without cirrhosis.
- Substudy 1, Arm B: DB Placebo: DB placebo QD for 12 weeks in participants without cirrhosis
- Substudy 1, Arm B: OL 2-DAA: OL 150 mg ABT-450/100 mg ritonavir/25 mg ABT-267 (2-DAA) QD for 12 weeks in participants without cirrhosis
Arm/Group | Substudy 1, Arm A: DB 2-DAA | Substudy 1, Arm B: DB Placebo | Substudy 1, Arm B: OL 2-DAA | Substudy 2, Arm C: OL 2-DAA
Serious Adverse Events (participants affected / at risk) | 7/215 | 2/106 | 3/106 | 2/42
Other Adverse Events (participants affected / at risk) | 116/215 | 48/106 | 47/106 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 1, Arm A: DB 2-DAA (N=215) | Substudy 1, Arm B: DB Placebo (N=106) | Substudy 1, Arm B: OL 2-DAA (N=106) | Substudy 2, Arm C: OL 2-DAA (N=42)
NECROTISING RETINITIS (Eye disorders) | 0 | 0 | 1 | 0
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 | 0 | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
GASTRIC CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
MULTIPLE SCLEROSIS (Nervous system disorders) | 1 | 0 | 0 | 0
ANURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 1, Arm A: DB 2-DAA (N=215) | Substudy 1, Arm B: DB Placebo (N=106) | Substudy 1, Arm B: OL 2-DAA (N=106) | Substudy 2, Arm C: OL 2-DAA (N=42)
ANAEMIA (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1
EYE DISCHARGE (Eye disorders) | 0 | 0 | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 4 | 0 | 3 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 0 | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 2 | 2 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 8 | 3 | 5 | 1
GLOSSODYNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 9 | 4 | 1 | 3
STOMATITIS (Gastrointestinal disorders) | 6 | 3 | 3 | 0
VOMITING (Gastrointestinal disorders) | 2 | 2 | 1 | 2
FACE OEDEMA (General disorders) | 2 | 0 | 0 | 1
FATIGUE (General disorders) | 6 | 1 | 1 | 1
FEELING HOT (General disorders) | 0 | 0 | 0 | 1
LOCAL SWELLING (General disorders) | 0 | 0 | 0 | 1
MALAISE (General disorders) | 9 | 3 | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 11 | 0 | 4 | 3
PYREXIA (General disorders) | 4 | 1 | 1 | 4
THIRST (General disorders) | 0 | 0 | 0 | 1
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 2 | 4 | 2 | 1
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 36 | 14 | 8 | 6
PHARYNGITIS (Infections and infestations) | 1 | 1 | 3 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 2 | 3 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0 | 3 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1 | 1
ALPHA-2 MACROGLOBULIN INCREASED (Investigations) | 0 | 0 | 0 | 1
APOLIPOPROTEIN A-I DECREASED (Investigations) | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 1 | 1
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0 | 0 | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 0 | 1 | 2
HAEMATOCRIT DECREASED (Investigations) | 1 | 0 | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 2 | 0 | 1 | 2
LYMPHOCYTE MORPHOLOGY ABNORMAL (Investigations) | 0 | 0 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 3
RED BLOOD CELL COUNT DECREASED (Investigations) | 2 | 0 | 0 | 1
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 | 1 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 2 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 0
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
DIZZINESS (Nervous system disorders) | 6 | 2 | 0 | 2
HEADACHE (Nervous system disorders) | 19 | 10 | 7 | 3
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 3 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 4 | 2 | 1 | 2
SPUTUM RETENTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 2
DERMAL CYST (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 3
ECZEMA ASTEATOTIC (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 10 | 4 | 4 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
RASH (Skin and subcutaneous tissue disorders) | 4 | 2 | 4 | 2
HYPERTENSION (Vascular disorders) | 2 | 2 | 1 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.